CLINICAL TRIAL: NCT04981730
Title: The Development and Evaluation of a Web-based Childbirth and Parenting Intervention Program: A Randomized Controlled Trial
Brief Title: The Development and Evaluation of a Web-based Childbirth and Parenting Intervention Program
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Medical University (Other)
Responsible Party: Principal Investigator, Shu Yu Kuo, Principal investigator, Taipei Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: N202103092
Record Dates: First submitted 2021-07-08; First posted 2021-07-29 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Parenting; Self Efficacy; Psychological Distress
Keywords: parenting; parenthood; web-based intervention; self-efficacy; psychological distress; infant health

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Web-based intervention (Experimental): Participants in the intervention will receive both the standardized usual care and guided web-based, individually-tailored childbirth and parenting intervention program, consisting of training sessions plus weekly email, message, or video-conference contact from their assigned nurse specialist.
  Interventions: Behavioral: Web-based intervention
- Control (No Intervention): Participants in the control group will receive attention from the research nurse and the standardized usual care.

INTERVENTIONS:
Behavioral: Web-based intervention — The web-based intervention participants will follow the website's orientation, the curriculum of modules, and professional feedback to complete the intervention.
  Arms: Web-based intervention

SUMMARY:
Background: The transition to parenthood is stressful for first-time mothers and fathers and links to adverse health outcomes. Despite Internet use's popularity, an effective web-based, individually-tailored intervention to enhance parental self-efficacy and infant health for first-time parents remains lacking.

Objectives: This study aims to develop and evaluate the effectiveness of a web-based, individually-tailored childbirth and parenting intervention program on parenting self-efficacy and infant health outcomes. The feasibility and acceptability of a theory-driven intervention will be examined in first-time mothers and fathers.

Methods: A two-arm, single-blind randomized controlled trial will be conducted to investigate the effects of web-based intervention in the first-time mother and father. Participants will be randomly allocated to a web-based intervention or a control condition. A repeated measurement will be performed.

Anticipatory results: The efficacy of a theory-driven web-based, individually tailored intervention program will provide a valuable contribution to perinatal health care for first-time mothers and fathers.

DETAILED DESCRIPTION:
The primary outcome of parenting self-efficacy and breastfeeding self-efficacy. The secondary outcomes of anxiety, depression, sleep quality, social support, infant health outcomes will be assessed. Data will be analyzed with the intention-to-treat analysis using linear mixed-effects modeling.

ELIGIBILITY:
Inclusion Criteria: for this study are first-time mothers and fathers who are

1. 20 years old and above;
2. primipara with a singleton pregnancy at second and third-trimester gestation;
3. able to read and write in Mandarin;
4. the husband or support partner will be willing to attend the intervention program;
5. able to access and use the Internet by computer and/or smartphone daily.

Exclusion Criteria: are the first-time mothers and fathers who have

1. chronic diseases;
2. obstetric complications;
3. an abnormal fetal screening;
4. unable or unwilling to comply with the requirements of the research protocol;
5. women and their partners did not have time for the web-based intervention program;
6. participation on any other interventional study.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 600 (Estimated)
Dates: Start 2023-12-14 (Actual); Primary Completion 2025-10-14 (Estimated); Study Completion 2025-10-14 (Estimated)

PRIMARY OUTCOMES:
Parenting self-efficacy | Baseline
  Parenting self-efficacy will be measured and reported by Parenting Self-Efficacy Scale. The higher the total scores indicate greater perceived parental self-efficacy.
Breastfeeding self-efficacy | Baseline
  Breastfeeding self-efficacy was measured using the Taiwanese version of the Maternal Breastfeeding Self-Efficacy Scale-Short Form (BSES-SF) and Breastfeeding self-efficacy Scale-Short Form among fathers (BSES-SFF). Total scores range from 14 to 70, with higher scores representing a higher level of self-efficacy.
Parenting self-efficacy | the third trimester of pregnancy
  Parenting self-efficacy will be measured and reported by Parenting Self-Efficacy Scale. The higher the total scores indicate greater perceived parental self-efficacy.
Breastfeeding self-efficacy | the third trimester of pregnancy
  Breastfeeding self-efficacy was measured using the Taiwanese version of the Maternal Breastfeeding Self-Efficacy Scale-Short Form (BSES-SF) and Breastfeeding self-efficacy Scale-Short Form among fathers (BSES-SFF). Total scores range from 14 to 70, with higher scores representing a higher level of self-efficacy.
Parenting self-efficacy | 1-month postpartum
  Parenting self-efficacy will be measured and reported by Parenting Self-Efficacy Scale. The higher the total scores indicate greater perceived parental self-efficacy.
Breastfeeding self-efficacy | 1-month postpartum
  Breastfeeding self-efficacy was measured using the Taiwanese version of the Maternal Breastfeeding Self-Efficacy Scale-Short Form (BSES-SF) and Breastfeeding self-efficacy Scale-Short Form among fathers (BSES-SFF). Total scores range from 14 to 70, with higher scores representing a higher level of self-efficacy.
Parenting self-efficacy | 3-month postpartum
  Parenting self-efficacy will be measured and reported by Parenting Self-Efficacy Scale. The higher the total scores indicate greater perceived parental self-efficacy.
Breastfeeding self-efficacy | 3-month postpartum
  Breastfeeding self-efficacy was measured using the Taiwanese version of the Maternal Breastfeeding Self-Efficacy Scale-Short Form (BSES-SF) and Breastfeeding self-efficacy Scale-Short Form among fathers (BSES-SFF). Total scores range from 14 to 70, with higher scores representing a higher level of self-efficacy.

SECONDARY OUTCOMES:
Depressive symptoms | Baseline, the third trimester of pregnancy,1-month postpartum and 3-month postpartum
  Depressive symptoms will be measured using the Taiwanese version of the Edinburgh Postnatal Depression Scale (T-EPDS). Total scores range from 0 to 30, A higher score indicated a higher levels of depression, with a total score of 30.
Anxiety symptoms | Baseline, the third trimester of pregnancy,1-month postpartum and 3-month postpartum
  Anxiety symptoms will be measured using the Taiwanese version of the State-Trait Anxiety Inventory (TSTAI). Total scores range from 20 to 80, with a high score indicating a high level of anxiety.
Sleep quality | Baseline, the third trimester of pregnancy,1-month postpartum and 3-month postpartum
  Sleep quality and disturbance will be measured using the Chinese version Pittsburgh Sleep Quality Index (CPSQI). CPSQI is a self-reported questionnaire and assesses seven sleep quality components from 0 to 3, with a total score ranging from 0 (good sleep) to 21 (very poor sleep).
Social support | Baseline, the third trimester of pregnancy,1-month postpartum and 3-month postpartum
  Social support will be measured using the Chinese version of the multidimensional scale of perceived social support (MSPSS). The higher the score, the higher the degree of support; total score ranging from 12 to 84.
Infant feeding methods | Baseline, the third trimester of pregnancy,1-month postpartum and 3-month postpartum
  Infant feeding methods will be measured using a self-report questionnaire. The feeding methods, including initiated breastfeeding within 24h after birth, and type of breastfeeding.
Infant sleep quality | 1-month postpartum and 3-month postpartum
  The infant sleep quality will be measured using the Taiwanese version of the Brief Infant Sleep Questionnaire (BISQ). The BISQ will be used to assess sleep duration, duration of sleep by circadian rhythm, and night-time awakenings.
Infant development | 3-month postpartum
  Infant development will be measured using the Taipei City Developmental Checklist for the assessment of developmental delay.
Feasibility measured using a structured questionnaire | immediately after intervention
  The feasibility of this trial will be measured using a structured questionnaire.
Satisfaction measured using a structured questionnaire | immediately after intervention
  Participants' satisfaction will be measured using a structured questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Shu-Yu Kuo, Principal Investigator — Taipei Medical University
Locations (1):
- Taipei Medical University Hospital, Taipei, Taiwan